CLINICAL TRIAL: NCT04004052
Title: Conservative Treatment Versus Ultrasound Guided Injection in Management of Meralgia Paresthetica: A Randomized Controlled Trial
Brief Title: Conservative Treatment and Ultrasound Guided Injection for Treatment Meralgia Paresthetica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ozturk84
Record Dates: First submitted 2019-05-17; First posted 2019-07-01 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Meralgia Paresthetica
Keywords: Meralgia paresthetica; Ultrasound-guided injection; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Femoral Neuropathy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Blockade of the LFCN is performed for therapeutic management of MP in group 1.
  Interventions: Other: Ultrasound guided injection
- Group 2 (Active Comparator): Ten sessions of conventional TENS were applied to the group 2 daily 20 minutes per session, 5 days per week, for 2 weeks.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS)
- Group 3 (Sham Comparator): Sham TENS was applied to the group 3 with the same protocol.
  Interventions: Other: Sham Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Other: Ultrasound guided injection
  Arms: Group 1
Other: Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: Group 2
Other: Sham Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: Group 3

SUMMARY:
Meralgia paresthetica (MP) is an entrapment mononeuropathy of the lateral femoral cutaneous nerve (LFCN), where conservative treatment options are not always sufficient.

The aim of this study was to evaluate the efficacy of ultrasound (US) guided lateral femoral cutaneous nerve injection in the management of meralgia paresthetica by comparing with transcutaneous electrical nerve stimulation (TENS) therapy and sham transcutaneous electrical nerve stimulation therapy.

DETAILED DESCRIPTION:
In this prospective, randomized, sham-controlled study, fifty four patients (23 female and 31 male, the mean age 53.61±11.99 years) with lateral femoral cutaneous nerve compression with clinical and electrophysiological findings were enrolled. Patients were randomly assigned to three groups: 1) Ultrasound-guided injection group, 2) TENS group, 3) Sham TENS group. The blockage of the lateral femoral cutaneous nerve was performed for therapeutic meralgia paresthetica management in group 1. Ten sessions of conventional TENS were administered to each patient 5 days a week for 2 weeks, for 20 minutes per daily session in Group 2, and sham TENS was applied to group 3 with the same protocol.

Visual Analog Scale (VAS), painDETECT questionnaire (PD-Q), Semmes Weinstein monofilament test (SWMt), Pittsburgh Sleep Quality Index (PSQI) and health-related quality of life (SF 36), at onset (T1), 15 days after treatment (T2) and 1 month after treatment (T3) were used for evaluation.

ELIGIBILITY:
Inclusion criteria

* Patients diagnosed with LFCN entrapment confirmed by clinical and electrophysiological findings

Exclusion criteria

* Secondary entrapment neuropathy
* Malignancy
* Pregnancy
* Infection in the inguinal region or dermatitis
* Lumbar radiculopathy
* Cardiac pacemakers
* Polyneuropathy

Ages: 42 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 months
  The VAS was used to record each patient's current level of pain with 0 indicating no pain and 10 indicating the worst pain that the patient had ever experienced. Using a ruler marked in centimeters, the examiner obtained the exact values along a 10-cm VAS line.
painDETECT questionnaire | 1 months
  It consists of seven items evaluating pain qualities, one evaluating the course of pain, and one evaluating pain radiation. Additionally, the questionnaire contains three numerical rating scales (NRSs) of 0-10 for current, worst, and average pain severity. An overall score is generated that summarizes everything but the pain intensity NRS, which ranges between -1 and 38. An overall score of >18 indicates likely Neuropathic pain, 13-18 possible Neuropathic pain, and < 13 unlikely Neuropathic pain.
Semmes-Weinstein monofilament test | 1 months
  Cutaneous pressure threshold was measured by touch test using a device with nylon Semmes-Weinstein monofilaments (SWMt) embedded in a plastic handle. A small pushing force is applied anterolateral femoral skin area for 1-1,5 seconds to push the filaments. A medical staff member presses the filaments at an angle of approximately 90° against the patient's thigh. This test is useful for medical staff because it is simple and easy. The threshold was defined as the lightest filament that the subject responses correctly at least two out of the three trials. The filaments are labeled with a numerical marking, which is a log to the base ten of the force in tenth of milligrams. Applications was made where the most symptoms has been observed in the patient's anterolateral thigh.

SECONDARY OUTCOMES:
Short Form (SF-36) Health Questionnaire | 1 months
  Assessment of health-related quality of life Health status was measured using the 36-Item Short Form (SF-36) Health Survey, version 2 (SF-36v2), which assesses eight different aspects of health. Item scores can be aggregated into physical component (PC) summary and mental component (MC) summary score.
Pittsburgh Sleep Quality Index (PSQI) | 1 Months
  PSQI is a 19-item self-reported instrument designed to measure a person's sleep quality and sleep patterns over 1-month time interval. It consists of seven items evaluating sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The 7 component scores are evaluated between 0 and 3 points. 3 reflects the negative extreme on the Likert Scale. The global score ranges from 0 to 21 points. Higher scores indicate worst sleep quality. A global score of >5 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Öztürk, MD, Principal Investigator — Fatih Sultan Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
This was a prospective, randomized, sham controlled study. Patients were randomly distributed into three groups: 1)US-guided injection group, 2)TENS group, 3)Sham TENS group. Blockade of the LFCN is performed for therapeutic management of MP in group 1. Ten sessions of conventional TENS were applied to the group 2 daily 20 minutes per session, 5 days per week, for 2 weeks while sham TENS was applied to the group 3 with the same protocol. Visual Analog Scale (VAS), painDETECT score, The Semmes-Weinstein monofilaments test (SWMt), The Pittsburgh Sleep Quality Index (PSQI), and assessment of health-related quality of life (SF 36) were used for evaluation at baseline (T1), post-treatment 15ᵗʰ day (T2), and 1st month post-treatment (T3).